CLINICAL TRIAL: NCT02792478
Title: Determination of RAS Mutation Status in Liquid Biopsies in Subjects With RAS Wild-type Colorectal Cancer in First-line Treatment: a Prospective, Observational Multi-centre Study in Spain. PERSEIDA Study
Brief Title: Determination of RAS Mutation Status in Liquid Biopsies in Subjects With RAS Wild-type.PERSEIDA Study
Acronym: PERSEIDA
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20140381
Record Dates: First submitted 2016-04-26; First posted 2016-06-07 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: RAS Wild Type mCRC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood samples will be collected according to the site's routine clinical practice usually prior to each treatment cycle and at the follow-up visits. Analysis of the RAS mutation status will be carried out on blood samples taken at baseline, on those carried out at 20 +/-2 weeks after the start of treatment (in any case, prior to the second tumour assessment) and on the sample obtained upon progression, coinciding with routine clinical practices for collecting blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RAS wild-type subjects: The blood samples will be collected according to the site's routine clinical practice usually prior to each treatment cycle and at the follow-up visits. Analysis of the RAS mutation status will be carried out on blood samples taken at baseline, on those carried out at 20 +/-2 weeks after the start of treatment (in any case, prior to the second tumour assessment) and on the sample obtained upon progression, coinciding with routine clinical practices for collecting blood. Blood Samples will be collected to all subjects participating (119 subjects.)Objective to evaluate the RAS mutation status at baseline in liquid biopsies in subjects with RAS wild type metastatic colorectal cancer.
- Patient RAS WT: As in cohort 1 blood samples will be collected for all subjects participating (119) 10 ml will be used for analysis of the RAS mutation status. The mutation status of BRAF and EGFR will be also analysed with the IdyllaTM (Biocartis) tests in this Cohort 2. In 20 patients included in Cohort 2, 10 ml additional taken at baseline will be used in order to determine the RAS mutation status by the BEAMing technique and 10 ml additional taken at disease progression will be used to determine the mutational profile in genes other than RAS by a NGS technique.

SUMMARY:
Analysis of freely circulating DNA in liquid biopsies using the BEAMing method

DETAILED DESCRIPTION:
Analysis of freely circulating DNA in liquid biopsies using the BEAMing method is proposed as a technique that may be useful for analysing the RAS mutation status in different types of cancer. However, first it is necessary to evaluate the concordance between the results obtained in tumour samples and liquid biopsies.

Primary objective

• To evaluate the RAS mutation status at baseline in liquid biopsies in subjects with RAS wild-type metastatic colorectal cancer.

Secondary objectives

* To evaluate the appearance of new RAS mutations using liquid biopsies at the moment of disease progression.
* To evaluate the appearance of new RAS mutations using liquid biopsies prior to radiological documentation of disease progression.

ELIGIBILITY:
Inclusion criteria:

* Subjects who give their informed consent in writing
* Subjects with metastatic colorectal cancer, measurable by RECIST, who start first-line treatment
* Male and female subjects, at least 18 years of age and of any ethnicity
* Subjects with a histologically-confirmed diagnosis of colorectal carcinoma with metastatic disease and wild-type RAS.

Exclusion criteria:

* Pregnant or breastfeeding women
* Subjects who have previously received monoclonal antibodies against EGFR (cetuximab or panitumumab), small-molecule EGFR inhibitors (such as erlotinib) or other biological cancer treatments
* History of another solid or haematological tumour in the previous 5 years, except a history of basal cell carcinoma of the skin or pre-invasive cervical cancer
* Subjects who are participating or have participated in a clinical trial in the 30 days prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with metastatic colorectal cancer, measurable by RECIST, who start first-line treatment
Sampling Method: Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Detection rate of RAS mutations in liquid biopsies in subjects with RAS wild-type mCRC at baseline. | Baseline
  To evaluate the RAS mutation status at baseline in liquid biopsies in two cohorts of subjects with RAS wild-type metastatic colorectal cancer: one analysed with the BEAMing (Sysmex-Inostics) technique (Cohort 1) and the other one analysed with the IdyllaTM (Biocartis) tests (Cohort 2).

SECONDARY OUTCOMES:
Description of RAS mutations using liquid biopsies at the moment of disease progression | Median time to progression ranges from 12 to 24 months
  Serial protocol specified radiographic and clinical assessment until disease progression
  One (plasma DNA) liquid biopsy performed at the time progression is documented.
  Progression time cannot be determined in advance of it's occurrence.
Description of the RAS mutations using liquid biopsies at 20 +/-2 weeks after starting treatment and prior to the second radiological assessment of the disease. | at 20+/- 2 weeks after treatment start
  The percentage of subjects who present RAS mutations in liquid biopsies taken prior to the second disease assessment will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (19):
- Spain (19):
  - Research Site, Almería, Andalusia
  - Research Site, Granada, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, San Cristóbal de La Laguna, Canary Islands
  - Research Site, Burgos, Castille and León
  - Research Site, Salamanca, Castille and León
  - Research Site, Lleida, Catalonia
  - Research Site, Terrassa, Catalonia
  - Research Site, Cáceres, Extremadura
  - Research Site, Ourense, Galicia
  - Research Site, Cartagena, Murcia
  - Research Site, Avilés, Principality of Asturias
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Alicante, Valencia
  - Research Site, Castellon, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
  - Research Site, Murcia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Valladares-Ayerbes M, Safont MJ, Gonzalez Flores E, Garcia-Alfonso P, Aranda E, Munoz AL, Falco Ferrer E, Cirera Nogueras L, Rodriguez-Salas N, Aparicio J, Llanos Munoz M, Pimentel Caceres PP, Castillo Trujillo OA, Vidal Tocino R, Salgado Fernandez M, Salud-Salvia A, Massuti Sureda B, Garcia-Carbonero R, Vicente Conesa MA, Lloansi Vila A; PERSEIDA investigators. Sequential RAS mutations evaluation in cell-free DNA of patients with tissue RAS wild-type metastatic colorectal cancer: the PERSEIDA (Cohort 2) study. Clin Transl Oncol. 2024 Oct;26(10):2640-2651. doi: 10.1007/s12094-024-03487-4. Epub 2024 Apr 20. PMID 38642257
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com